CLINICAL TRIAL: NCT05884450
Title: The Effect of Acupressure on the Management of Dyspnea in Palliative Care Patients
Brief Title: The Effect of Acupressure on the Management of Dyspnea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul Aydın University (Other)
Responsible Party: Principal Investigator, DİLEK YILDIRIM, Principal Investigator, Istanbul Aydın University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ACUPRESSURE DYSPNEA
Record Dates: First submitted 2023-05-08; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Palliative Care; Dyspnea
Keywords: Acupressure; Palliative Care; Dyspnea; Nursing
MeSH Terms: conditions — Dyspnea | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment (Experimental): In the experimental group, acupressure will be applied to the patients by the researchers twice a day, every day for two weeks, for 3 minutes to each point (Lu1, Lu10, P6).
  Interventions: Other: Acupressure
- Control (No Intervention): No application will be made to the control group.

INTERVENTIONS:
Other: Acupressure — Acupressure is an integrated method of applying physical pressure to acupuncture points on the body surface with hands, elbows or various tools. With good counseling, patients can apply this method, which is non-invasive, easy to apply and safe, on their own.
  Arms: Experiment

SUMMARY:
Dyspnea can develop at any stage of the disease, but it is more common in the last period of life.

Complementary and integrative methods used for dyspnea symptoms include acupuncture, acupressure, visualization techniques, herbal treatments, nutritional supplements, stress management, relaxation techniques, exercise, breathing training and psychotherapy, etc. There are studies in the literature showing that acupuncture and acupressure are effective in controlling dyspnea symptoms in various disease groups.

Acupressure is an integrated method of applying physical pressure to acupuncture points on the body surface with hands, elbows or various tools. With good counseling, patients can apply this method, which is non-invasive, easy to apply, and safe.

Reducing the psychological stress that causes dyspnea along with dyspnea is important for symptom management. It has been reported that acupressure application has significant effects especially in dyspnea that develops with exertion. It is seen that studies on the subject are not sufficient in terms of quantity and quality in terms of giving advice to patients, and there is a need for well-planned studies with high power.

The aim of this study; The aim of this study is to determine the effect of acupressure applied to three acupuncture points (Lu1, Lu10, P6) on the arm and chest in palliative care patients with dyspnea on dyspnea level and quality of life, twice a day for 4 weeks, for 3 minutes to each point.

DETAILED DESCRIPTION:
Dyspnea can develop at any stage of the disease, but it is more common in the last period of life (1). In different studies, the incidence of dyspnea in patients receiving palliative care with the diagnosis of lung cancer was reported to be 57-90%, 60% in esophageal cancer, and 46% in breast cancer (1-5). In a study, it was shown that 65% of palliative care patients died with dyspnea in the last three months of their lives (6). There may be many reasons that trigger the development of dyspnea in palliative care patients. In addition to primary or metastatic lung involvement, antineoplastic therapy, thoracic irradiation, obstruction caused by mediastinal tumor, pleural effusion and pulmonary embolism may also cause dyspnea. In addition, dyspnea in these patients may be due to existing chronic obstructive pulmonary disease, pulmonary embolism, hepatomegaly, acidity, anemia that can affect the patient's respiration, cachexia, anxiety, or thoracic surgery (7). Regardless of the cause, as a result, dyspnea is one of the important complaints that negatively affects the patient's quality of life and reminds patients of death. Since dyspnea is a multifaceted subjective condition that affects the patient physiologically, psychologically, socially and environmentally, comprehensive diagnosis and early planning of effective approaches in its management are important for patients to complete a good palliative care process (8-10).

Complementary and integrative methods used for dyspnea symptoms include acupuncture, acupressure, visualization techniques, herbal treatments, nutritional supplements, stress management, relaxation techniques, exercise, breathing training and psychotherapy, etc. (11,12) There are studies in the literature showing that acupuncture and acupressure are effective in controlling dyspnea symptoms in various disease groups (13,14).

Acupressure is an integrated method of applying physical pressure to acupuncture points on the body surface with hands, elbows or various tools. With good counseling, patients can apply this method, which is non-invasive, easy to apply, and safe (13).

Reducing the psychological stress that causes dyspnea along with dyspnea is important for symptom management (10). It has been reported that acupressure application has significant effects especially in dyspnea that develops with exertion (14). It is seen that studies on the subject are not sufficient in terms of quantity and quality in terms of giving advice to patients, and there is a need for well-planned studies with high power.

The aim of this study; The aim of this study is to determine the effect of acupressure applied to three acupuncture points (Lu1, Lu10, P6) on the arm and chest in palliative care patients with dyspnea on dyspnea level and quality of life, twice a day for 4 weeks, for 3 minutes to each point.

Method:

Purpose and Type of Study: The aim of the study, which will be conducted in randomized controlled parallel group, experimental research design type, is to determine the effect of acupressure on dyspnea level and quality of life in palliative care patients with dyspnea symptoms.

Variables of the Study Independent Variable: Socioeconomic and disease-related characteristics (age, gender, diagnosis, length of hospital stay, etc.).

Dependent Variable: Quality of Life, level of dyspnea, vital signs. Intervention to be Implemented In the experimental group, acupressure will be applied to the patients by the researchers twice a day, every day for two weeks, for 3 minutes to each point (Lu1, Lu10, P6). No application will be made to the control group. Respiratory rate, rhythm, blood pressure, heart rate and Borg Scale Score will be evaluated and recorded for 14 days before and after acupressure application. On the 7th and 14th days, the FACIT - Pal (Functional Assessment of Chronic Illness Therapy- Palliative care) Quality of Life Scale will be filled again.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older,
* Least literate,
* Patients with moderate to severe dyspnea (with dyspnea score of 3 or higher on a 0-10 scale in the Modified Borg Scale evaluation) will be included in the study.

Exclusion Criteria:

* Refusal to participate in the study
* Finding a communication problem

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-05-22 (Estimated); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Patient Descriptive Information Form: | Baseline
  In the form prepared by the researchers; There are 20 questions about the personal characteristics of the patients and the disease, palliative care and dyspnea.
Modified Borg Scale (MBS) | Baseline
  The first version of the MBS was developed in 1970 by Gunnar Borg to measure the effort expended during physical exercise. The scale was rearranged in 1982 and turned into a scale consisting of 12 items diagnosing the severity of dyspnea according to their degrees (15). As the scores on the scale increase, the severity of dyspnea increases.
Change Modified Borg Scale (MBS) | 2nd day
  The first version of the MBS was developed in 1970 by Gunnar Borg to measure the effort expended during physical exercise. The scale was rearranged in 1982 and turned into a scale consisting of 12 items diagnosing the severity of dyspnea according to their degrees (15). As the scores on the scale increase, the severity of dyspnea increases.
Change Modified Borg Scale (MBS) | 3th day
  The first version of the MBS was developed in 1970 by Gunnar Borg to measure the effort expended during physical exercise. The scale was rearranged in 1982 and turned into a scale consisting of 12 items diagnosing the severity of dyspnea according to their degrees (15). As the scores on the scale increase, the severity of dyspnea increases.
Change Modified Borg Scale (MBS) | 4th day
  The first version of the MBS was developed in 1970 by Gunnar Borg to measure the effort expended during physical exercise. The scale was rearranged in 1982 and turned into a scale consisting of 12 items diagnosing the severity of dyspnea according to their degrees (15). As the scores on the scale increase, the severity of dyspnea increases.
Change Modified Borg Scale (MBS) | 5th day
  The first version of the MBS was developed in 1970 by Gunnar Borg to measure the effort expended during physical exercise. The scale was rearranged in 1982 and turned into a scale consisting of 12 items diagnosing the severity of dyspnea according to their degrees (15). As the scores on the scale increase, the severity of dyspnea increases.
Change Modified Borg Scale (MBS) | 6th day
  The first version of the MBS was developed in 1970 by Gunnar Borg to measure the effort expended during physical exercise. The scale was rearranged in 1982 and turned into a scale consisting of 12 items diagnosing the severity of dyspnea according to their degrees (15). As the scores on the scale increase, the severity of dyspnea increases.
Change Modified Borg Scale (MBS) | 7th day
  The first version of the MBS was developed in 1970 by Gunnar Borg to measure the effort expended during physical exercise. The scale was rearranged in 1982 and turned into a scale consisting of 12 items diagnosing the severity of dyspnea according to their degrees (15). As the scores on the scale increase, the severity of dyspnea increases.
Change Modified Borg Scale (MBS) | 8th day
  The first version of the MBS was developed in 1970 by Gunnar Borg to measure the effort expended during physical exercise. The scale was rearranged in 1982 and turned into a scale consisting of 12 items diagnosing the severity of dyspnea according to their degrees (15). As the scores on the scale increase, the severity of dyspnea increases.
Change Modified Borg Scale (MBS) | 9th day
  The first version of the MBS was developed in 1970 by Gunnar Borg to measure the effort expended during physical exercise. The scale was rearranged in 1982 and turned into a scale consisting of 12 items diagnosing the severity of dyspnea according to their degrees (15). As the scores on the scale increase, the severity of dyspnea increases.
Change Modified Borg Scale (MBS) | 10th day
  The first version of the MBS was developed in 1970 by Gunnar Borg to measure the effort expended during physical exercise. The scale was rearranged in 1982 and turned into a scale consisting of 12 items diagnosing the severity of dyspnea according to their degrees (15). As the scores on the scale increase, the severity of dyspnea increases.
Change Modified Borg Scale (MBS) | 11th day
  The first version of the MBS was developed in 1970 by Gunnar Borg to measure the effort expended during physical exercise. The scale was rearranged in 1982 and turned into a scale consisting of 12 items diagnosing the severity of dyspnea according to their degrees (15). As the scores on the scale increase, the severity of dyspnea increases.
Change Modified Borg Scale (MBS) | 12th day
  The first version of the MBS was developed in 1970 by Gunnar Borg to measure the effort expended during physical exercise. The scale was rearranged in 1982 and turned into a scale consisting of 12 items diagnosing the severity of dyspnea according to their degrees (15). As the scores on the scale increase, the severity of dyspnea increases.
Change Modified Borg Scale (MBS) | 13th day
  The first version of the MBS was developed in 1970 by Gunnar Borg to measure the effort expended during physical exercise. The scale was rearranged in 1982 and turned into a scale consisting of 12 items diagnosing the severity of dyspnea according to their degrees (15). As the scores on the scale increase, the severity of dyspnea increases.
Change Modified Borg Scale (MBS) | 14th day
  The first version of the MBS was developed in 1970 by Gunnar Borg to measure the effort expended during physical exercise. The scale was rearranged in 1982 and turned into a scale consisting of 12 items diagnosing the severity of dyspnea according to their degrees (15). As the scores on the scale increase, the severity of dyspnea increases.
Functional Assessment of Chronic Illness Therapy- Palliative Care (FACIT - Pal) | Baseline
  The validity and reliability of the scale, which was developed by David Cella et al. in 1993 (16) with palliative care patients, was performed by Lyons et al. in 2009 (17). This assessment tool, which is used to evaluate the quality of life of palliative care patients, consists of a total of 46 statements and 5 sub-dimensions. High scores obtained from the total of the scale indicate high quality of life, and low scores indicate a decrease in quality of life.
Change Functional Assessment of Chronic Illness Therapy- Palliative Care (FACIT - Pal) | 7th Day
  The validity and reliability of the scale, which was developed by David Cella et al. in 1993 (16) with palliative care patients, was performed by Lyons et al. in 2009 (17). This assessment tool, which is used to evaluate the quality of life of palliative care patients, consists of a total of 46 statements and 5 sub-dimensions. High scores obtained from the total of the scale indicate high quality of life, and low scores indicate a decrease in quality of life.
Change Functional Assessment of Chronic Illness Therapy- Palliative Care (FACIT - Pal) | 14th Day
  The validity and reliability of the scale, which was developed by David Cella et al. in 1993 (16) with palliative care patients, was performed by Lyons et al. in 2009 (17). This assessment tool, which is used to evaluate the quality of life of palliative care patients, consists of a total of 46 statements and 5 sub-dimensions. High scores obtained from the total of the scale indicate high quality of life, and low scores indicate a decrease in quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Dilek Yildirim, Istanbul, Küçükçekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided